CLINICAL TRIAL: NCT06252350
Title: Clinical Evaluation of Radiation Reduction for Optimized Safety - Pilot Study
Brief Title: CERROS Pilot Study
Acronym: CERROS - Pilot
Status: Completed | Type: Observational
Sponsor: Angiowave Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-PLAN-101v1
Record Dates: First submitted 2024-02-02; First posted 2024-02-09 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Coronary Disease; Coronary Stenosis; Angina Pectoris; Chest Pain
Keywords: CAD; Coronary; Angina; PCI; Angiography
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Coronary Disease; Coronary Stenosis; Angina Pectoris; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to determine whether a reduced radiation protocol (RRP) in which angiograms are acquired at ultralow radiation doses and then processed using spatiotemporal enhancement software can produce similar quality angiographic images as compared with standard techniques.

DETAILED DESCRIPTION:
Coronary angiography is an essential diagnostic tool for determining the presence and severity of coronary artery disease, a leading cause of morbidity and mortality worldwide. While the basic techniques of coronary angiography have remained unchanged, the field of medical imaging has undergone significant advancements in hardware and software, offering new possibilities for enhanced visualization of the coronary arteries, better diagnostic accuracy, and improved patient and staff safety. However, the use of radiation during coronary angiography, which is necessary for image acquisition, exposes patients, physicians, and staff to potential risks, including radiation-induced tissue damage and an increased long-term risk of cancer. While the risks to patients attributable to the relatively low radiation doses they receive during single catheterization procedures are minimal, the cumulative risks of occupational radiation exposure are higher among physicians and staff, who are repetitively exposed to scattered radiation on a daily basis and accumulated over the course of years working in the catheterization laboratory. This occupational radiation exposure has been associated with an increased risk of cataracts, premature atherosclerosis, and certain cancers among physicians and staff. There is therefore a pressing need to explore strategies to minimize radiation doses used during coronary angiography without compromising the diagnostic accuracy of coronary artery disease detection.

Recent advancements in computational power and image processing algorithms provide opportunities for substantial reductions in radiation doses used during coronary angiography. One such advancement is spatiotemporal enhancement processing (STEP) which improves the signal to noise ratio of time sequenced angiographic data and enhances the visibility of vascular structure. This innovative STEP technique has the promise of minimizing patient and operator radiation exposure while maintaining adequate image quality. The purpose of this pilot study is to investigate a novel strategy of radiation dose reduction and data processing in coronary angiography. This pilot study will be performed in patients undergoing clinically-indicated diagnostic coronary angiography.

The study will compare angiograms acquired at ultralow radiation doses and processed with spatiotemporal enhancement software (STEP-angiograms) to standard of care angiograms (SOC-angiograms) acquired with normal radiation dose settings and no additional processing. The objectives are to assess offline whether the low radiation STEP-angiograms are of equivalent diagnostic quality as SOC-angiograms. In future research studies, the STEP software will be tested in the clinical setting to evaluate how the software may improve patient safety, enhance the overall quality of care, promote the responsible use of radiation in coronary angiography procedures, and reduce occupational radiation doses among physician and staff in the catheterization laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Referred for clinically indicated coronary angiography
* ≥18 years of age
* Not pregnant
* English speaking
* Not imprisoned
* Able to provide written informed consent

Exclusion Criteria:

* Hemodynamically or electrically unstable.
* Indication for coronary angiography is emergent, including ST-segment elevation myocardial infarction
* History of coronary artery bypass grafting
* An eGFR <60
* Pregnant or lactating
* A BMI of 45 or greater
* Any other factor that the investigator feels would put the patient at increased risk or otherwise make the patient unsuitable for participation in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected to have coronary artery disease (CAD) who are undergoing diagnostic coronary angiography with or without possible percutaneous coronary intervention (PCI).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Segment-level percent diameter stenosis (%DS) | Periprocedural
  Segment-level quantitative coronary angiography (QCA) determination of percent diameter stenosis (%DS)

SECONDARY OUTCOMES:
Stenosis severity | Periprocedural
  Agreement in reader-adjudication of segment-level identification of mild/intermediate/severe stenosis
Diagnostic quality | Periprocedural
  Percent of coronary segments qualitatively determined to be of adequate diagnostic image quality
Radiation dose - SOC | Periprocedural
  Radiation dose (air kerma and dose-area product) for SOC-angiograms
Radiation dose - STEP | Periprocedural
  Radiation dose (air kerma and dose-area product) for STEP-angiograms

CONTACTS AND LOCATIONS:
Overall Officials: Ryan D Madder, MD, Principal Investigator — Corewell Health; Sean P Madden, PhD, Study Director — Angiowave Imaging; Aram Salzman, Study Chair — Angiowave Imaging
Locations (1):
- Corewell Health West, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months
URL: http://www.angiowaveimaging.com

REFERENCES:
- [Background] Ryan TJ. The coronary angiogram and its seminal contributions to cardiovascular medicine over five decades. Circulation. 2002 Aug 6;106(6):752-6. doi: 10.1161/01.cir.0000024109.12658.d4. No abstract available. PMID 12163439
- [Background] The 2007 Recommendations of the International Commission on Radiological Protection. ICRP publication 103. Ann ICRP. 2007;37(2-4):1-332. doi: 10.1016/j.icrp.2007.10.003. PMID 18082557
- [Background] Valentin J. Avoidance of radiation injuries from medical interventional procedures. Ann ICRP. 2000;30(2):7-67. doi: 10.1016/S0146-6453(01)00004-5. PMID 11459599
- [Background] Andreassi MG, Cioppa A, Botto N, Joksic G, Manfredi S, Federici C, Ostojic M, Rubino P, Picano E. Somatic DNA damage in interventional cardiologists: a case-control study. FASEB J. 2005 Jun;19(8):998-9. doi: 10.1096/fj.04-3287fje. Epub 2005 Mar 31. PMID 15802491
- [Background] Karatasakis A, Brilakis HS, Danek BA, Karacsonyi J, Martinez-Parachini JR, Nguyen-Trong PJ, Alame AJ, Roesle MK, Rangan BV, Rosenfield K, Mehran R, Mahmud E, Chambers CE, Banerjee S, Brilakis ES. Radiation-associated lens changes in the cardiac catheterization laboratory: Results from the IC-CATARACT (CATaracts Attributed to RAdiation in the CaTh lab) study. Catheter Cardiovasc Interv. 2018 Mar 1;91(4):647-654. doi: 10.1002/ccd.27173. Epub 2017 Jul 14. PMID 28707381